CLINICAL TRIAL: NCT07038668
Title: The Innovative Appliance of Cohesive Viscoelastic During Pars Plana Vitrectomy in Complicated Ocular Trauma
Status: Not yet recruiting | Type: Observational
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xueying Zhongliu, Clinical Professor, Zhongshan Ophthalmic Center, Sun Yat-sen University
Other Study IDs: 2025KYPJ043
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Ocular Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposed Group
  Interventions: Procedure: Using of viscoelastic during the operation
- Non-Exposed Group
  Interventions: Procedure: No using of viscoelastic during the operation

INTERVENTIONS:
Procedure: Using of viscoelastic during the operation — Using of viscoelastic during the operation
  Groups: Exposed Group
Procedure: No using of viscoelastic during the operation — No using of viscoelastic during the operation
  Groups: Non-Exposed Group

SUMMARY:
Viscoelastic is a powerful tool in pars plana vitrectomy(PPV) surgery relative to perfluorocarbon liquid because it has the properties to dilate and engorge the retina and restore the detached retina to its original position. We intend to explore whether the use of viscoelastic to assist PPV surgery can help improve surgical efficiency, reduce tissue damage, and improve the outcomes of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Severe traumatic ocular injury (ocular trauma score, OTS=1 or 2)
* PVR retinal detachment (Stage D2 or D3)

Exclusion Criteria:

* Visual acuity below the base line before injury

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will be selected from the outpatient department of Zhongshan Ophthalmic Center
Sampling Method: Non-Probability Sample
Enrollment: 420 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Best Corrected Visual Acuity(BCVA) | From enrollment to the end of follow up in 3 months
  Best Corrected Visual Acuity
Reattachment of Retina | Post operation till the end of follow up in 3 months
  Check through ultrasound, optical coherence tomography(OCT) to see if retina is reattached.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol